CLINICAL TRIAL: NCT04893720
Title: The SPINUS II Study: Spinal Fusion for Multilevel SPECT/CT Positive Lumbar Degeneration
Status: Recruiting | Type: Observational
Sponsor: Military University Hospital, Prague (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Radek Kaiser, Principal Investigator, Military University Hospital, Prague
Other Study IDs: SPINUS-UVN II
Record Dates: First submitted 2021-05-15; First posted 2021-05-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Disc Disease; Back Pain Lower Back Chronic; Facet Joint Arthropathy; Facet Syndrome of Lumbar Spine
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lumbar fusion — Transforaminal Lumbar Interbody Fusion of the SPECT/CT positive lumbar degeneration

SUMMARY:
The aim of the present study is to find out whether fusion of multilevel SPECT/CT positive lumbar degeneration leads to a significant improvement of pain and disability.

DETAILED DESCRIPTION:
Chronic back pain (CBP) is a very common clinical problem. It is dominantly caused by degenerative changes, while specific causes such as tumor, trauma or inflammatory conditions are relatively rare. Back pain may be a concomitant symptom of lumbar disc herniation or spinal canal stenosis and is a typical symptom of spondylolisthesis. Magnetic resonance imaging (MRI) plays a key role in the diagnosis, showing in detail the soft structures, vertebral bodies (Modic changes, MC) or signs of facet arthropathy. On the other hand, it also proves a number of clinically silent findings. Degenerative disc disease (DDD) or facet osteoarthritis are most often considered to be a pain generator. The problem, however, is that both entities are very common in the general population without a painful correlate, and there is still controversy in the literature about their role in the genesis of CBP.

Radionuclide bone scintigraphy with single photon emission computed tomography (SPECT) provides functional imaging and is used to detect microcalcification due to increased osteoblastic activity. In the absence of other pathology the foci of increased osteoblastic activity reflex areas of mechanical stress and degenerative change in the skeleton. There is growing evidence about the relationship between DDD, facet arthropathy, and SPECT positivity. Although these findings have been recently confirmed by surgical studies, the evidence about the effect of surgical treatment of SPECT positive lumbar degeneration is still weak due to the small number of operated patients.

The aim of the present study is to define a possible correlation between degenerative changes of the lumbar spine and positivity on SPECT/CT imaging. Patients with multilevel SPECT+ DDD or facet arthropathy will undergo spinal fusion of the involved segments. Postoperative improvement will be measured by ODI (Oswestry Disability Index) and pain VAS (Visual Analogue Scale) in 6 and 24 months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Lower back pain (in extension +/- pain in buttocks, groin, thigh) without radicular pain
* Symptoms > 6 months after the failure of conservative management in the primary care setting
* MRI signs of degenerative disc disease or facet arthropathy
* Two- or more levels of positivity on lumbar SPECT/CT

Exclusion Criteria:

* Other spinal pathology (tumors, congenital defects, spondylolysis, or spondylolisthesis)
* Intolerance of SPECT examination
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An open prospective cohort study will be performed. Inclusion criteria will be: subjects between 18 and 75 years of age; both genders; with CBP and diagnosis of DDD or facet arthropathy on MRI and increased metabolic activity on bone SPECT/CT imaging in the same levels who are undergoing open lumbar interbody fusion. New MRI of the lumbar spine and SPECT/CT will be performed 2 years after the surgical procedure. The patients will complete ODI and VAS questionnaires before surgery and at 6- and 24-months follow-up visits. All patients will sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | 2 years
  The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. he scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Change in Pain Visual Analogue Scale (VAS) | 2 years
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between VAS 0 (no pain) and VAS 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslav Plas, Study Chair — jaroslav.plas@uvn.cz
Locations (2):
- Czechia (2):
  - Military University Hospital Prague, Prague
  - University Hospital, Motol, Prague

IPD SHARING:
Plan to Share IPD: No